CLINICAL TRIAL: NCT04464525
Title: Omecamtiv Mecarbil Post-trial Access Protocol for Subjects Completing Study 20110203 GALACTIC-HF
Brief Title: Omecamtiv Mecarbil Post-trial Access Study
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20190370
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Chronic Heart Failure With Reduced Ejection Fraction
MeSH Terms: interventions — omecamtiv mecarbil

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Omecamtiv mecarbil (Experimental): All subjects will be assigned to OM
  Interventions: Drug: Omecamtiv mecarbil

INTERVENTIONS:
Drug: Omecamtiv mecarbil — Film-coated tablet administered orally.
  Other Names: AMG 423

SUMMARY:
The primary objective of this study is to provide access to omecamtiv mecarbil for participants who have completed GALACTIC-HF 20110203.

DETAILED DESCRIPTION:
This study was conducted by Amgen as the IND holder, with Cytokinetics as a collaborator. Due to the termination of the collaboration agreement between Amgen and Cytokinetics in May 2021 and subsequent transfer of the omecamtiv mecarbil IND from Amgen to Cytokinetics, Cytokinetics is now listed as the sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided GALACTIC-HF PTA informed consent prior to initiation of any study specific activities/procedures.
* Participant has completed GALACTIC-HF.

Exclusion Criteria:

* Investigational product was permanently discontinued during GALACTIC-HF due to protocol-specified reason.
* Female participant is pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 5 days after the last dose of treatment.
* Female participants of childbearing potential unwilling to use 2 acceptable methods of effective contraception during treatment with OM and for an additional 5 days after the last dose of treatment.
* Female participants of childbearing potential with a positive pregnancy test assessed on day 1 by a urine pregnancy test.
* Participant has known sensitivity to any of the products or components to be administered during dosing.
* History or evidence of any clinically significant disorder, condition or disease that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to participant safety or interfere with the study evaluation, procedures or completion.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-18 (Estimated); Primary Completion 2026-11-27 (Estimated); Study Completion 2026-11-27 (Estimated)

PRIMARY OUTCOMES:
Number of participants administered omecamtiv mecarbil during the treatment period | Up to 252 weeks
  Primary analysis is based on the exploratory outcome measure.

OTHER OUTCOMES:
Participant incidence of serious adverse events and treatment emergent adverse events | Up to 252 weeks
  Targeted adverse events are those which lead to temporary or permanent discontinuation of OM, adverse events that are possibly related to OM or study procedures, and all adverse events of myocardial infarction, myorcardial ischemia, and ventricular arrhythmia, irrespective of seriousness and relationship to OM.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com